CLINICAL TRIAL: NCT05414175
Title: A Phase 3, Open-label, Single Arm, Clinical Study to Evaluate Efficacy, Safety and Tolerability of Mavacamten in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study of Mavacamten in Obstructive Hypertrophic Cardiomyopathy
Acronym: HORIZON-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV027-004
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiomyopathy, Hypertrophic Obstructive
Keywords: Mavacamten; Obstructive Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mavacamten (Experimental)
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: BMS-986427; MYK-461

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and tolerability of a 30-week course of mavacamten and the long-term effects of mavacamten in Japanese participants with symptomatic obstructive hypertrophic cardiomyopathy (HCM).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and greater, body weight ≥ 35kg
* Has adequate acoustic windows to enable accurate transthoracic echocardiograms (TTEs)
* Diagnosed with obstructive hypertrophic cardiomyopathy consistent with current American College of Cardiology Foundation/American Heart Association, European Society of Cardiology, and Japanese Circulation Society guidelines
* Has documented left ventricular ejection fraction (LVEF) ≥60% NYHA Class II or III

Exclusion Criteria:

* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics oHCM, such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to Screening
* History of resuscitated sudden cardiac arrest (at any time) or known history of appropriate implantable cardioverter defibrillator (ICD) discharge for life-threatening ventricular arrhythmia within 6 months prior to Screening
* Paroxysmal atrial fibrillation with atrial fibrillation present at the time of Screening.
* Persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to Screening and/or not adequately rate controlled within 6 months prior to Screening
* Treatment (within 14 days prior to Screening) or planned treatment during the study with cibenzoline, disopyramide or ranolazine
* Treatment (within 14 days prior to Screening) or planned treatment during the study with a combination of beta blockers and verapamil or a combination of beta blockers and diltiazem
* Has been successfully treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to Screening or plans to have either of these treatments during the study
* ICD placement within 2 months prior to Screening or planned ICD placement during the study
* Has a history or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation procedures, or completion
* Prior treatment with cardiotoxic agents such as doxorubicin or similar

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2025-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- Japan (20):
  - Local Institution - 0020, Uwajima, Ehime
  - Local Institution - 0026, Himeji-Shi, Hyōgo
  - Local Institution - 0016, Kobe, Hyōgo
  - Local Institution - 0017, Tsukuba, Ibaraki
  - Local Institution - 0023, Kanazawa, Ishikawa-ken
  - Local Institution - 0019, Yokohama, Kanagawa
  - Local Institution - 0015, Nankoku-shi, Kochi
  - Local Institution - 0028, Tsu, Mie-ken
  - Local Institution - 0027, Sendai, Miyagi
  - Local Institution - 0014, Suita, Osaka
  - Local Institution - 0011, Suita-Shi, Osaka
  - Local Institution - 0012, Hamamatsu, Shizuoka
  - Local Institution - 0010, Bunkyo-Ku, Tokyo
  - Local Institution - 0009, Chuo-Ku, Tokyo
  - Local Institution - 0003, Fuchu-Shi, Tokyo
  - Local Institution - 0001, Itabashi-Ku, Tokyo
  - Local Institution - 0007, Koto-Ku, Tokyo
  - Local Institution - 0005, Shinjuku-Ku, Tokyo
  - Local Institution - 0013, Shinjuku-ku, Tokyo
  - Local Institution - 0018, Osaka

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Mavacamten: Participants with symptomatic obstructive hypertrophic cardiomyopathy received oral capsule of mavacamten during the treatment period from Day 1 to Week 30. The starting dose of mavacamten was 2.5 milligram (mg) once daily. At Week 6, Week 8, Week 14, and Week 20, mavacamten dose were titrated based on the individual, transthoracic echocardiogram (TTE) response (Valsalva left ventricular outflow tract [LVOT] gradient and left ventricular ejection fraction LVEF). The permissible doses during the study were 1, 2.5, 5, 10, or 15 mg.
Period: Overall Study
Arm/Group | Mavacamten
Started | 38
Intent to Treat Population (All participants who passed screening or assigned study drug.) | 38
Safety Population (All participants who receive at least one dose of study drug.) | 38
Completed | 36
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mavacamten
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-exercise Left Ventricular Outflow Tract (LVOT) Peak Gradient at Week 30
Description: The post-exercise LVOT gradient was measured from echocardiograms obtained at baseline and week 30 following a study-specified exercise protocol and read by the doppler echocardiography. Baseline is defined as the last non-missing assessment prior to the first dose of the study treatment if both the time of the measurement and the time of first dose are available otherwise it is the last non-missing assessment on or prior to the first dose of the study treatment.
Time Frame: At Baseline and Week 30
Population: Intent-to-treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Mavacamten
Number analyzed (Participants) | 35
millimeters of mercury (mmHg) | -60.6963 (31.55674)

2. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire 23-item Version (KCCQ-23) Clinical Summary Score (CSS) at Week 30
Description: The KCCQ-23 is a 23-item, self-administered questionnaire that measures the impact of a participant's cardiovascular disease or its treatment on 6 distinct domains using a 2-week recall period: symptoms/signs, physical limitation, quality of life (QoL), social limitations, self-efficacy, and symptom stability. The KCCQ 23 Clinical Summary Score (CSS) is derived from the Total Symptom Score (TSS) and the Physical Limitations (PL) score of the KCCQ 23. The CSS, TSS, and the PL score range from 0 to 100 with higher scores representing less severe symptoms and/or physical limitations. The CSS is a mean of the TSS and the PL score. Baseline is defined as the last non-missing assessment prior to the first dose of the study treatment if both the time of the measurement and the time of first dose are available otherwise it is the last non-missing assessment on or prior to the first dose of the study treatment.
Time Frame: At Baseline and Week 30
Population: Intent to Treat Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Mavacamten
Number analyzed (Participants) | 36
Score on a Scale | 9.766 (16.8588)

3. Secondary Outcome: Percentage of Participants With at Least 1 Class Improvement in New York Heart Association (NYHA) Functional Class From Baseline to Week 30
Description: The NYHA Functional Classification of Heart Failure (HF) assigns participants to 1 of 4 categories based on the participant's symptoms. Class I (No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea); Class II (Slight limitation of physical activity, Comfortable at rest, Ordinary physical activity results in fatigue, palpitation, dyspnea); Class III (Marked limitation of physical activity, Comfortable at rest, Less-than ordinary-activity causes fatigue, palpitation, or dyspnea) and Class IV (Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases). Improvement is defined as participant moving to lower class category from a higher one. Baseline is defined as last non-missing measurement prior to the first dose.
Time Frame: Baseline and at Week 30
Population: Intent To Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Mavacamten
Number analyzed (Participants) | 38
Percentage of participants | 63.2

4. Secondary Outcome: Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Week 30
Description: Blood samples were collected for assessing the concentration of NT-proBNP. Baseline is defined as last non-missing measurement prior to the first dose.
Time Frame: At baseline and week 30
Population: Intent to Treat Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: nanogram per liter (ng/L)
Arm/Group | Mavacamten
Number analyzed (Participants) | 36
nanogram per liter (ng/L) | -738.0 [-3101 to 590]

5. Secondary Outcome: Change From Baseline in Cardiac Troponin I at Week 30
Description: Blood samples were collected for assessing cardiac troponins. Baseline is defined as the last non-missing assessment prior to the first dose of the study treatment if both the time of the measurement and the time of first dose are available otherwise it is the last non-missing assessment on or prior to the first dose of the study treatment.
Time Frame: At baseline and week 30
Population: Intent to Treat population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Mavacamten
Number analyzed (Participants) | 36
ng/L | -10.920 [-226.42 to 0.80]

6. Secondary Outcome: Change From Baseline in Cardiac Troponin T at Week 30
Description: as for outcome 5
Time Frame: At baseline and week 30
Population: Intent to Treat Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Mavacamten
Number analyzed (Participants) | 36
ng/L | -4.95 [-19.2 to 0.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality was measured from first dose up until approximately 66 weeks post-first dose. SAEs and Other AEs were collected from first dose till last dose plus 140 days (up to approximately 50 weeks).
Description: Safety analysis population included all participants who receive at least one dose of study drug.
Arm/Group | Mavacamten
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 6/38
Other Adverse Events (participants affected / at risk) | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=38)
Atrial fibrillation (Cardiac disorders) | 1
Macular oedema (Eye disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=38)
Atrial fibrillation (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 2
Cataract (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Malaise (General disorders) | 2
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT05414175/Prot_SAP_000.pdf